CLINICAL TRIAL: NCT00271726
Title: Prospective, Randomized, Multi-Center Pilot Study on the Treatment of Unstable, Extraarticular Colles Fractures of the Distal Radius by Palmar Locking Plate, External Fixator or Kirschner Wires
Brief Title: Operative Treatment of Extraarticular Colles' Fractures of the Distal Radius (OTEC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Philipps University Marburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTEC Pilot 1 KKS MR
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Colles' Fracture; Radius Fractures
Keywords: distal radius fracture; extraarticular Colles fracture
MeSH Terms: conditions — Colles' Fracture; Radius Fractures; Wrist Fractures | interventions — Fracture Fixation, Internal; External Fixators; Bone Wires

INTERVENTIONS:
Procedure: Osteosynthesis with palmar locking plate
Procedure: Osteosynthesis with external fixator
Procedure: Osteosynthesis with Kirschner wires

SUMMARY:
This is a prospective, randomized, multi-center pilot study of unstable extraarticular fractures of the distal radius with dorsal displacement of the distal fragment in elderly patients. The patients are randomly assigned to osteosynthesis with palmar locking plate, external fixator, or Kirschner wires.

The aim of this pilot study is to allow a sample size calculation for a main randomized controlled trial (RCT). The primary outcome criterion is the functional status measured by the Disability of the Arm, Shoulder and Hand (DASH) questionnaire. Secondary outcome criteria are pain, range of motion (ROM), grip strength, and radiological parameters. Since this is a pilot study it is intended to generate a study hypothesis for the main RCT.

ELIGIBILITY:
Inclusion Criteria:

* Isolated, extraarticular, unstable Colles' fracture of the metaphysis of the distal radius (AO type A3)
* Age 65 years or older
* Patient agreed with and signed the "informed consent" form

Exclusion Criteria:

* Fractures older than 7 days (more than 1 week between injury and treatment)
* Other injuries of the hand
* Other relevant injuries of the upper extremities
* Open fracture
* Patients with one hand missing
* Clinical or radiological signs of any rheumatoid disease, osteoarthritis, or polyarthritis
* Previous skeletal injury or severe soft tissue injury of the arm
* History of drug or alcohol abuse
* Patients unlikely to cooperate or attend all scheduled visits
* Patients who have participated in any other device or drug clinical trial within the previous month
* Patients with legal incompetence

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90
Dates: Start 2005-11

PRIMARY OUTCOMES:
Functional status measured by DASH questionnaire

SECONDARY OUTCOMES:
Pain
Range of motion (ROM)
Grip strength
Radiological parameters
Feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schädel-Höpfner, MD, Principal Investigator — Department of Trauma and Hand Surgery, University Hospital, Moorenstrasse 5, D - 40225 Düsseldorf
Locations (1):
- Department of Trauma and Hand Surgery, University Hospital, Düsseldorf, Germany